CLINICAL TRIAL: NCT01909934
Title: A Phase 4, Open-label, Single-Arm Study of Brentuximab Vedotin in Patients With Relapsed or Refractory Systemic Anaplastic Large Cell Lymphoma
Brief Title: Study of Brentuximab Vedotin in Participants With Relapsed or Refractory Systemic Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25006; 2012-004128-39 (EudraCT Number); U1111-1154-9784 (Registry Identifier: WHO); REec-2014-0649 (Registry Identifier: REec); 13/NI/0072 (Registry Identifier: NRES)
Record Dates: First submitted 2013-07-01; First posted 2013-07-29 (Estimated); Results first posted 2022-05-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
Keywords: Lymphoma; Anaplastic Large-cell; Relapsed; Refractory; Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; monomethyl auristatin E; Drug Therapy; Immunotherapy; Hematologic Diseases
MeSH Terms: conditions — Lymphoma; Recurrence; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Anaplastic; Hematologic Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin 1.8 mg/kg (Experimental): Participants received brentuximab vedotin 1.8 mg/kg as a 30 minute intravenous (IV) infusion on Day 1 of each 3 week cycle. Participants with stable disease or better and without unacceptable toxicity were to receive a minimum of 8 cycles with the opportunity to receive a maximum of 16 cycles.
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Brentuximab vedotin IV infusion
  Other Names: SGN-35; ADCETRIS

SUMMARY:
The purpose of this study is to assess the antitumor efficacy of single-agent brentuximab vedotin 1.8 mg/kg administered intravenously (IV) every 3 weeks, as measured by the overall objective response rate (ORR) in patients with r/r sALCL following at least 1 multiagent chemotherapy regimen (cyclophosphamide, doxorubicin hydrochloride [hydroxydaunorubicin], vincristine sulfate [Oncovin], and prednisone [CHOP] or equivalent multiagent chemotherapy regimens with curative intent).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants age 18 years or older, with relapsed or refractory sALCL who have previously received at least 1 multiagent chemotherapy
* Bidimensional measurable disease
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Female participants who are postmenopausal for at least 1 year before the screening visit, surgically sterile, or agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 30 days after the last dose of study drug, or agree to practice true abstinence
* Male participants who agree to practice effective barrier contraception during the entire study treatment period through 6 months after the last dose of study drug or agree to practice true abstinence
* Clinical laboratory values as specified in the study protocol

Exclusion Criteria:

* Previous treatment with brentuximab vedotin.
* Previously received an allogeneic transplant.
* Participants with current diagnosis of primary cutaneous anaplastic large cell lymphoma [ALCL] (participants whose ALCL has transformed to sALCL are eligible).
* Known cerebral/meningeal disease including signs or symptoms of progressive multifocal leukoencephalopathy (PML)
* Female participants who are lactating and breastfeeding or pregnant
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (40):
- Belgium (4):
  - ZNA Stuivenberg, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Croatia (3):
  - Clinical Hospital Centre Rijeka, Rijeka
  - Clinical Hospital Centre Zagreb, Zagreb
  - Clinical Hospital Dubrava, Zagreb
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem, Pécs
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Malopolskie Centrum Medyczne s.c., Krakow
  - SPZOZ MSW zWarminsko-MazurskimCen.Onko.wOlsztynie, Olsztyn
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
- Portugal (4):
  - Hospital de Braga, Braga
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto, E.P.E. - Hospital de Santo Antonio, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (4):
  - Policlinica de Diagnostic Rapid SA, Brasov
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
- Spain (5):
  - ICO lHospitalet Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Turkey (Türkiye) (6):
  - Ankara University Medical Faculty, Ankara
  - Pamukkale Uni. Med. Fac., Denizli
  - Istanbul Bilim University Medical Fac., Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Erciyes University Medical Faculty, Kayseri
- United Kingdom (3):
  - Royal Cornwall Hospital, Truro, Cornwall
  - The Christie, Manchester, Greater Manchester
  - Birmingham Heartlands Hospital, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 23 January 2014 to 29 August 2024.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory systemic anaplastic large cell lymphoma were enrolled to receive brentuximab vedotin 1.8 milligrams per kilogram (mg/kg).
Period: Overall Study
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Started | 50
Completed | 19
Not Completed | 31
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Death | 25
Not completed — Withdrawal of Informed Consent | 1
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least 1 dose of brentuximab vedotin.
Groups:
- Brentuximab Vedotin 1.8 mg/kg: Participants received brentuximab vedotin 1.8 mg/kg as a 30 minute IV infusion on Day 1 of each 3 week cycle. Participants with stable disease or better and without unacceptable toxicity were to receive a minimum of 8 cycles with the opportunity to receive a maximum of 16 cycles.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (16.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1
  Croatia | 2
  Czech Republic | 12
  Hungary | 5
  Poland | 8
  Portugal | 3
  Romania | 3
  Spain | 4
  Turkey | 6
  United Kingdom | 6
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 166.8 (10.40)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 75.2 (20.73)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] — BMI= weight/height^2, where weight is in kilograms and height in meters.
  kilograms per meter squared (kg/m^2) | 26.9 (6.39)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a complete remission (CR) or partial remission (PR) by Independent Review Facility (IRF) response assessment according to the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma. CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites.
Time Frame: Up to data cut-off date: 04 May 2021 (Up to approximately 7 years)
Population: Intent-to-Treat Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
percentage of participants | 64 [49 to 77]

2. Secondary Outcome: Duration of Response (DOR) Per IRF
Description: DOR was defined as the time between initial response and documented tumor progression in the subset of participants who achieved an objective response, either CR or PR. DOR per IRF was based upon the radiological assessment of measured lesions from an independent review facility. DOR was censored on the date of the last disease assessment documenting absence of progressive disease (PD) for participants who were lost to follow-up, withdrew consent, started a new anticancer therapy other than stem cell transplant (SCT), or discontinued treatment due to undocumented PD after the last adequate disease assessment.
Time Frame: Until disease progression, death, or the data cut-off date: 4 May 2021 (Up to approximately 7 years)
Population: Intent-to-Treat Population included all participants enrolled in the study. Only responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 32
months | NA [19.71 to NA] — Median and upper limit of confidence interval (CI) were not estimable as most of the responders were censored.

3. Secondary Outcome: Progression-free Survival (PFS) Per IRF
Description: PFS is defined as the time from start of study treatment to first documentation of objective tumor progression or to death due to any cause, whichever comes first. PFS per IRF is based upon the radiological assessment from an independent review facility.
Time Frame: Until disease progression, death, or the data cut-off date: 4 May 2021 (Up to approximately 7 years)
Population: Intent-to-Treat Population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
months | 20.9 [4.17 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events up to data cut-off date: 4 May 2021.

4. Secondary Outcome: Complete Remission Rate (CRR) Per IRF
Description: CRR is defined as percentage of participants with CR. CR is defined as the disappearance of all evidence of disease.
Time Frame: Until disease progression, death, or the data cut-off date: 4 May 2021 (Up to approximately 7 years)
Population: Intent-to-Treat Population included all participants enrolled in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
percentage of participants | 30 [18 to 45]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from start of study treatment to date of death due to any cause.
Time Frame: Until disease progression, death, or end of study (Up to approximately 10.7 years)
Population: Intent-to-Treat Population included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
months | 67.6 [17.68 to NA] — Upper limit of 95% CI was not estimable due to insufficient number of participants with events.

6. Secondary Outcome: Percentage of Participants Receiving Hematopoietic Stem Cell Transplant (SCT) Following Treatment With Brentuximab Vedotin
Time Frame: Until disease progression, death, or end of study (Up to approximately 10.7 years)
Population: Intent-to-Treat Population included all participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
percentage of participants | 28

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs and TEAEs by Severity (Grade 3 or Higher)
Description: An adverse event (AE): any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to medicinal product. TEAE was defined as any AE that started after the first administration of study drug in this continuation study. Serious TEAEs: defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect, or is a medically important event.
Time Frame: From first dose up to 30 days post last dose of study drug (Up to approximately 1 year)
Population: Safety Population included all participants who received at least 1 dose of brentuximab vedotin.
Measure: Number; unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
percentage of participants
  TEAEs | 94
  Serious TEAEs | 32
  Drug-Related TEAEs | 70
  TEAEs by Severity (Grade 3 or Higher) | 58

8. Secondary Outcome: Concentration of Serum Antibody-drug Conjugate (ADC) at the End of Infusion
Time Frame: Cycle 1, Day 1 and Cycle 3, Day 1 at the end of infusion
Population: Pharmacokinetic (PK) Population included participants who received at least 1 dose of brentuximab vedotin and have PK concentration data available. Number analyzed are participants with data available for analyses at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per liter (µg/L)
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
micrograms per liter (µg/L)
  Cycle 1, Day 1: number analyzed (Participants) | 48
  Cycle 1, Day 1 | 35 (35)
  Cycle 3, Day 1: number analyzed (Participants) | 38
  Cycle 3, Day 1 | 38 (25)

9. Secondary Outcome: Concentration of Serum Total Antibody (TAb) Conjugate Plus Free Total Antibody
Time Frame: Cycle 1, Day 1 and Cycle 3, Day 1 at the end of infusion
Population: PK Population included participants who received at least 1 dose of brentuximab vedotin and have PK concentration data available. Number analyzed are participants with data available for analyses at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
µg/L
  Cycle 1, Day 1: number analyzed (Participants) | 48
  Cycle 1, Day 1 | 33 (29)
  Cycle 3, Day 1: number analyzed (Participants) | 36
  Cycle 3, Day 1 | 38 (23)

10. Secondary Outcome: Maximum Concentration for Unconjugated Drug- Monomethyl Auristatin E (MMAE)
Time Frame: Cycle 1, Day 1 and Cycle 3, Day 1 at the end of infusion
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 50
nanogram per milliliter (ng/ml)
  Cycle 1, Day 1: number analyzed (Participants) | 49
  Cycle 1, Day 1 | 0.25 (87)
  Cycle 3, Day 1: number analyzed (Participants) | 38
  Cycle 3, Day 1 | 0.29 (88)

11. Secondary Outcome: Percentage of Participants With Presence of Anti-Therapeutic Antibodies (ATA) and Neutralizing Antibodies (NAb) to Brentuximab Vedotin
Time Frame: Up to 16 cycles (each cycle = 21 days)
Population: Immunogenicity-evaluable Population included all participants who received at least 1 dose of brentuximab vedotin and had a baseline and at least 1 post-baseline sample available for evaluation for the presence of ATA and NAb. Overall number analyzed are participants with data available for analyses at the given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
Number analyzed (Participants) | 44
percentage of participants
  ATA Positive | 30
  Neutralizing ATA Positive | 0.0

ADVERSE EVENTS:
Time Frame: All-cause mortality: Throughout the study (Up to approximately 10.7 years); Serious and other adverse events: From first dose up to 30 days post last dose of study drug (up to approximately 1 year)
Description: The Safety Population included all participants who received at least 1 dose of brentuximab vedotin.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg
All-Cause Mortality (participants affected / at risk) | 25/50
Serious Adverse Events (participants affected / at risk) | 16/50
Other Adverse Events (participants affected / at risk) | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg (N=50)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Aortic stenosis (Vascular disorders) | 1
Autonomic neuropathy (Nervous system disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Central nervous system haemorrhage (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epididymitis (Infections and infestations) | 1
General physical health deterioration (General disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ischaemic stroke (Nervous system disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg (N=50)
Anaemia (Blood and lymphatic system disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3
Malaise (General disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 8
Oedema peripheral (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 9
Pyrexia (General disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 4
Vomiting (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT01909934/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT01909934/SAP_001.pdf